CLINICAL TRIAL: NCT01002950
Title: Multicenter, Randomized, Double-Masked, Placebo-Controlled, Dose Escalation, Multiple-Dose Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of ACU-4429 in Subjects With Dry Age-Related Macular Degeneration (Geographic Atrophy)
Brief Title: Study of the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ACU-4429 in Subjects With Geographic Atrophy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kubota Vision Inc. (Industry)
Collaborators: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4429-201
Record Dates: First submitted 2009-10-26; First posted 2009-10-28 (Estimated); Last update posted 2014-03-11 (Estimated); Status verified 2014-02

CONDITIONS: Dry Age-related Macular Degeneration; Geographic Atrophy
MeSH Terms: conditions — Geographic Atrophy | interventions — emixustat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ACU-4429 tablet (Experimental)
  Interventions: Drug: ACU-4429
- Matching placebo tablet (Placebo Comparator)
  Interventions: Drug: Matching placebo

INTERVENTIONS:
Drug: ACU-4429 — ACU-4429 tablets (2, 5, 7, or 10 mg) taken orally once daily for 90 days
  Arms: ACU-4429 tablet
Drug: Matching placebo — Matching placebo tablets taken orally once daily for 90 days
  Arms: Matching placebo tablet

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of the investigational drug ACU-4429 in subjects with geographic atrophy.

ELIGIBILITY:
Inclusion Criteria:

* Have a clinical diagnosis of geographic atrophy, as defined in the protocol

Exclusion Criteria:

* Currently receiving or has received a medication prohibited by the protocol

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2009-10; Primary Completion 2012-06 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Safety as measured by: AEs, clinical laboratory tests, vital signs, physical exams, visual tests, and questionaire | Through treatment period (up to Day 90) until 1-2 weeks post last dose (Day 97-104)

SECONDARY OUTCOMES:
Pharmacokinetics as measured by plasma ACU-4429 drug levels | Baseline; Treatment Days 2, 7, 14, 30, 60 and 90

CONTACTS AND LOCATIONS:
Overall Officials: John W Chandler, MD, Study Director — Kubota Vision Inc.
Locations (12):
- United States (12):
  - Retinal Consultants of Arizona, Phoenix, Arizona
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - Covance Clinical Research Unit, Inc., Daytona Beach, Florida
  - National Ophthalmic Research Institute, Fort Meyers, Florida
  - Covance Clinical Research Unit, Inc., Honolulu, Hawaii
  - Kresege Eye Institute, Detroit, Michigan
  - Associated Retinal Consultants, P.C. / William Beaumont Hospital, Royal Oak, Michigan
  - New York Eye and Ear Infirmary, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Black Hills Regional Eye Institute, Rapid City, South Dakota
  - Covance Clinical Research Unit, Austin, Texas
  - Covance Clinical Research Unit, Inc., Dallas, Texas

REFERENCES:
- [Derived] Yeong JL, Loveman E, Colquitt JL, Royle P, Waugh N, Lois N. Visual cycle modulators versus placebo or observation for the prevention and treatment of geographic atrophy due to age-related macular degeneration. Cochrane Database Syst Rev. 2020 Dec 17;12(12):CD013154. doi: 10.1002/14651858.CD013154.pub2. PMID 33331670